CLINICAL TRIAL: NCT06620133
Title: The Effect of Pain Education and Patient-led Goal Setting Compared to Guideline-based Written Information on Pain and Disability in Adults With Chronic Low Back Pain: a Randomised Controlled Trial
Brief Title: Pain Education and Patient-led Goal Setting in Adults With Chronic Low Back Pain: a Randomised Controlled Trial
Acronym: CAPACITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroscience Research Australia (Other)
Responsible Party: Principal Investigator, Matthew Jones, Principal Investigator, Neuroscience Research Australia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPACITY trial
Record Dates: First submitted 2024-09-22; First posted 2024-10-01 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Chronic Low Back Pain (Non-specific, Uncomplicated)
Keywords: pain education; patient-led goal setting; chronic low back pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain education and patient-led goal setting (Experimental): Pain education and patient-led goal setting
  Interventions: Other: Pain education and patient-led goal setting
- Written advice (Experimental): Guideline-based written advice developed for people with chronic low back pain (e.g. https://pubmed.ncbi.nlm.nih.gov/34283182/)
  Interventions: Other: Guideline-based written advice

INTERVENTIONS:
Other: Pain education and patient-led goal setting — 8 week program delivered via five, up to 1-hour telehealth sessions. The sessions will be scheduled at approximately fortnightly intervals. Participants will also be prescribed approximately 30 minutes of online activities with each session. Pain education will be based on Explain Pain and the curriculum will have specified learning objectives adapted for each individual participant. Participants will access the online education curriculum through Pathwright. For patient-led goal setting, the healthcare practitioner will take an initial history of the participants physical activity behaviours and problems related to their back pain. The participant will prioritise their problems according to impact in their life. Strategies will then be discussed, and the participant will, in collaboration with the healthcare practitioner, set goals and strategies to work on independently between sessions.
  Arms: Pain education and patient-led goal setting
Other: Guideline-based written advice — Participants will receive guideline-based written information for the management of chronic low back pain. This will include information about the prognosis of low back pain and treatment options to consider.
  Arms: Written advice

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of two treatments for adults with chronic low back pain. The main question this study seeks to answer is "In adults with chronic low back pain, what is the effectiveness of pain education and patient-led goal setting compared to guideline-based written advice on reducing pain intensity and disability?".

A total of 392 participants will be randomised into two groups: 1) pain education and patient-led goal setting or 2) guideline-based written advice. Participants randomised to the pain education and patient-led goal setting group will receive 5 sessions of 45-60 min each over 8 weeks delivered online via telehealth. Participants randomised to written advice group will receive information developed for people with chronic low back pain. Outcomes will be assessed at baseline and week 8, 26 and 52.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain of at least 3 months duration
* physically inactive (less than or equal to 150min/week moderate intensity physical activity; 75 min/week vigorous activity, or some combination of the two)
* no known contraindication(s) to performing physical activity
* English language proficiency
* access to internet

Exclusion Criteria:

* physically active (more than 150min/week moderate intensity physical activity, 75 min/week vigorous activity, or some combination of the two)
* known contraindication(s) to performing physical activity
* known or suspected serious spinal pathology (fracture, metastatic, inflammatory or infective diseases of the spine, cauda equina syndrome/widespread neurological disorder)
* scheduled for major surgery during the treatment or follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2025-06-09 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Week 26 post-randomisation
  Average pain intensity over the previous 7 days assessed using the 11-point Numerical Pain Rating Scale
Disability | Week 26 post-randomisation
  Self-reported disability assessed using the Roland Morris Disability Questionnaire (RMDQ); scale range 0-24; lower scores indicate lower disability

SECONDARY OUTCOMES:
Pain intensity | Weeks 8 and 52 post-randomisation
  Average pain intensity over the previous 7 days assessed using the 11-point Numerical Pain Rating Scale
Disability | Weeks 8 and 52 post-randomisation
  Self-reported disability assessed using the Roland Morris Disability Questionnaire (RMDQ); scale range 0-24; lower scores indicate lower disability
Pain self-efficacy | Weeks 8, 26 and 52 post-randomisation
  Pain self-efficacy assessed using the Pain Self-Efficacy Questionnaire (PSEQ); scale range 0-60; higher scores indicate greater pain self-efficacy
Back beliefs | Weeks 8, 26 and 52 post-randomisation
  Back beliefs assessed using the Back Beliefs Questionnaire (BBQ); scale range 9-45, lower scores indicate more pessimistic beliefs about the consequences of low back pain
Kinesiophobia | Weeks 8, 26 and 52 post-randomisation
  Fear of movement (re)injury assessed by the short-form of the Tampa Scale of Kinesiophobia; scale range 4-16 (higher scores indicate greater kinesiophobia)
EuroQol 5-Dimension 5-Level (EQ-5D-5L) | Weeks 8, 26 and 52 post-randomisation
  Health-Related Quality of Life assessed using the EQ-5D-5L dimensions scale range, 1-5; higher scores indicate better quality of life) and health thermometer (range, 0-100; higher scores indicate better quality of life).
Daily step count | Week 8 post-randomisation
  Average daily step count over the past 7 days assessed using accelerometry.
Light intensity physical activity | Week 8 post-randomisation
  Light intensity physical activity (min/day) over the past 7 days assessed using accelerometry
Moderate-vigorous intensity physical activity | Week 8 post-randomisation
  Moderate-vigorous intensity physical activity (min/day) over the past 7 days assessed using accelerometry
Sedentary time | Week 8 post-randomisation
  Sedentary time (min/day) over the past 7 days assessed using accelerometry
Subjective physical activity levels | Weeks 8, 26 and 52 post-randomisation
  Self-reported physical activity over the previous 7 days assessed using the short-form of the International Physical Activity Questionnaire (IPAQ)
Lifestyle risk factors | Weeks 8, 26 and 52 post-randomisation
  Diet (do you eat less than two serves of fruit per day? (yes/no); do you eat less than fives serves of vegetables per day? (yes/no)).
  Alcohol intake (On average, how much alcohol do you drink each week? (I rarely/never drink alcohol; Less than 14 standard drinks; Between 14 and 21 standard drinks; More than 21 standard drinks)
Blood pressure | Week 8 post-randomisation
  Blood pressure at rest assessed via an automated sphygmomanometer
Adverse events | From randomisation to Week 8 post-randomisation
  Adverse events assessed via self-report
Adherence to treatment | From randomisation to Week 8 post-randomisation
  Adherence to treatment assessed via session attendance and self-report (diary)
Total healthcare costs | Weeks 8, 26 and 52 post-randomisation
  Total health-care costs will be estimated as the trial intervention costs and outside trial health-care resource use attributable to chronic low back pain from the Medicare Benefits Scheme and Pharmaceutical Benefits Scheme. Quality-adjusted life-years (QALYs) from the EQ-5D-5L using the Australian utility weights will also be used in the trial-based cost-utility analysis.
Goal attainment (goal setting arm only) | Weeks 8, 26 and 52 post-randomisation
  Goal attainment assessed using the goal attainment scale. Each goal is rated on a 5-point scale: +2 = much more than expected, +1 = somewhat more than expected, 0 = Patient achieves the expected level, -1 = somewhat less than expected, -2 = much less than expected.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Jones, Principal Investigator — UNSW Sydney
Locations (1):
- Neuroscience Research Australia, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made to interested researchers only upon reasonable request and once the proposed research project has received separate ethics approval from a Human Research Ethics Committee.
  Request to the data custodian, the Principal Investigator (matthew.jones@unsw.edu.au)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available after the publication of study reports. There is no end date for the availability of study data

REFERENCES:
- [Background] Gardner T, Refshauge K, McAuley J, Hubscher M, Goodall S, Smith L. Combined education and patient-led goal setting intervention reduced chronic low back pain disability and intensity at 12 months: a randomised controlled trial. Br J Sports Med. 2019 Nov;53(22):1424-1431. doi: 10.1136/bjsports-2018-100080. Epub 2019 Feb 26. PMID 30808666